CLINICAL TRIAL: NCT01419145
Title: A Feasibility Study of Multimodal Exercise/Nutrition/Anti-inflammatory Treatment for Cachexia - the Pre-MENAC Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: University of Edinburgh (Other); Oslo University Hospital (Other); NHS Greater Glasgow and Clyde (Other); Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010/2620 (REK); 2010-022897-14 (EudraCT Number)
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Cancer; Cachexia
Keywords: cachexia; neoplasms; complications; combined modality therapy; exercise therapy; diet therapy; anti-inflammatory agents
MeSH Terms: conditions — Neoplasms; Cachexia | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal intervention (Experimental)
  Interventions: Other: Multimodal intervention
- Standard Care (Active Comparator)
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Multimodal intervention — Nutritional supplements aimed at optimal energy balance and protein intake (2 cartons of ProSure per day), nutritional advice, home-based self-assisted exercise program and anti-inflammatory treatment (300 mg celecoxib) for 6 weeks. The aerobic exercise program is performed as self-administered daily walking sessions, aiming for a minimum of two sessions 30 minutes on a weekly basis. Other aerobic activities could be used instead of walking. The resistance exercise program should be performed 3 times weekly and lasts about 20 minutes. The program is targeting major muscle groups in the upper body and legs with use of weights. The intensity of the exercise and performance of the exercises are adapted to the individual patient's disease burden and physical performance.
  Arms: Multimodal intervention
Other: Standard care — Standard cancer care
  Arms: Standard Care

SUMMARY:
A multicentre, open, randomized phase II study comparing a multimodal intervention (oral nutritional supplements, celecoxib and physical exercise) for cachexia versus standard cancer care.

ELIGIBILITY:
Main eligibility criteria:

* Advanced non-small-cell lung cancer (stage III-IV) or pancreatic cancer not eligible for curative therapy
* Due to commence chemo- or chemo radiotherapy
* Karnofsky Performance Score ≥ 70
* A life expectancy of ≥4 months and considered able to complete 2 months of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-10; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment and retention | 12 weeks
  The aim of this study is to investigate the feasibility of the multimodal intervention for cancer cachexia by assessing; enrolment rate, compliance with study intervention, contamination-rate in the control group with respect to any of the interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Stein Kaasa, MD, PhD, Principal Investigator — National Taiwan Normal University; Ken Fearon, MD, PhD, Principal Investigator — University of Edinburgh
Locations (3):
- Norway (2):
  - Oslo University Hospital Ullevål, Oslo
  - St Olavs Hospital, Trondheim
- University of Edinburgh, Edinburgh, United Kingdom

REFERENCES:
- [Result] Solheim TS, Laird BJA, Balstad TR, Stene GB, Bye A, Johns N, Pettersen CH, Fallon M, Fayers P, Fearon K, Kaasa S. A randomized phase II feasibility trial of a multimodal intervention for the management of cachexia in lung and pancreatic cancer. J Cachexia Sarcopenia Muscle. 2017 Oct;8(5):778-788. doi: 10.1002/jcsm.12201. Epub 2017 Jun 14. PMID 28614627
- [Derived] Balstad TR, Brunelli C, Pettersen CH, Schonberg SA, Skorpen F, Fallon M, Kaasa S, Bye A, Laird BJA, Stene GB, Solheim TS. Power Comparisons and Clinical Meaning of Outcome Measures in Assessing Treatment Effect in Cancer Cachexia: Secondary Analysis From a Randomized Pilot Multimodal Intervention Trial. Front Nutr. 2021 Jan 14;7:602775. doi: 10.3389/fnut.2020.602775. eCollection 2020. PMID 33585533
- [Derived] Stene GB, Balstad TR, Leer ASM, Bye A, Kaasa S, Fallon M, Laird B, Maddocks M, Solheim TS. Deterioration in Muscle Mass and Physical Function Differs According to Weight Loss History in Cancer Cachexia. Cancers (Basel). 2019 Dec 3;11(12):1925. doi: 10.3390/cancers11121925. PMID 31816924